CLINICAL TRIAL: NCT01483794
Title: Genital Warts: Studies for Establishing Epidemiological Profile, Psychosocial Consequences and Costs of Disease in Attendants to the Sexual Health Clinic of the Public Health Service of Valparaiso and San Antonio, Chile.
Brief Title: Epidemiology, Costs and Psychosocial Consequences of Genital Warts in Valparaiso, Chile
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Carolina San Martin, Principal investigator, Universidad de Valparaiso
Other Study IDs: CondValpo2011; 1501 (Other: Servicio Salud Valparaiso-San Antonio Chile)
Record Dates: First submitted 2011-11-23; First posted 2011-12-01 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Condylomata Acuminata
Keywords: genital warts
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Genital warts treated: Patients that have had treatment on their genital warts
- Genital warts on treatment: Patients currently being treated for genital warts

SUMMARY:
This is an observational study looking at the characteristics of patients consulting for genital warts in the first semester 2010 at the public sexual health clinic of Valparaiso, Chile. The objectives are: to have an epidemiological profile, estimating cost of the disease for the health system and the patient and analyzing possible psychosocial consequences of the condition for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older
* Having being diagnosed with genital warts
* Consulting the sexual health clinic only for genital warts
* Patients accepting to be included in the study

Exclusion Criteria:

* Immunodeficiency
* HIV positive
* Having being diagnosed with cancer or pre-cancerous lesions
* Pregnancy
* Presenting a sexual transmissible infection other than genital warts.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the public sexual health clinic of Valparaiso, Chile
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with altered psychosocial tests as a Measure of impact of presenting genital warts. | one year
  The psychosocial consequences of presenting genital warts will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina San Martin, MD, Principal Investigator — University of Valparaiso, Chile
Locations (2):
- Chile (2):
  - Sexual Health Clinic,, Valparaíso, Región de Valparaíso
  - Sexual Health Clinic, Valparaíso, Región de Valparaíso